CLINICAL TRIAL: NCT03894579
Title: Phase 1, Open-Label, Safety Study of Escalating Doses of Ex Vivo Expanded, Autologous Natural Killer Cells in Subjects With Plaque Psoriasis
Brief Title: Autologous Natural Killer Cells in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNK01-MX03
Record Dates: First submitted 2019-03-06; First posted 2019-03-28 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Plaque Psoriasis
Keywords: natural killer cells; autologous

STUDY DESIGN:
Intervention Model Description: Non-randomized, open label, single center trial. Subjects will receive SNK01 using a 3 + 3 dose escalating design
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SNK01 (Experimental): SNK01 infused weekly for 4 consecutive weeks
  Interventions: Biological: Study Product: SNK01

INTERVENTIONS:
Biological: Study Product: SNK01 — SNK01 administered using an intravenous line (IV) to all patients at weeks 1, 2, 3, and 4

SUMMARY:
This is a non-randomized, dose escalating and open-labeled clinical trial to evaluate the safety of autologous natural killer cell (NK) infusions (IV) of "SNK01" in adults with plaque psoriasis. The primary objective of this study is to investigate the safety and tolerability of four infusions of "SNK01" in subjects with plaque psoriasis. Secondary objective is preliminary efficacy of "SNK01" in subjects with plaque psoriasis.

DETAILED DESCRIPTION:
Nine (9) subjects, male or female, aged 18 years or older will be enrolled in the study, all of whom will receive "SNK01" without placebo control. There are three (3) subjects in each of the three (3) cohorts. The SNK01 study product will be administered at the following doses using dose escalating rules: Cohort 1 will receive 4 weekly infusions of 1 billion cells, Cohort 2 will receive 4 weekly infusions of 2 billion cells, and Cohort 3 will receive 4 weekly infusions of 4 billion cells. Length of participation, per subject, is approximately 12 weeks. The primary endpoint for safety is dose-limiting toxicity (DLT) which is defined as TEAE of grade ≥ 3 considered related to SNK01. Secondary safety endpoints include other adverse events (graded according to National Cancer Institute's Common Toxicity Criteria for Adverse Events [NCI-CTCAE v 5.0]), vital sign measurements, clinical laboratory tests and physical examination. Preliminary efficacy will be measured by Psoriasis Area Severity Index (PASI) and by the Physician's Global Assessment (PGA.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered eligible for participation in the study if all the following inclusion criteria are satisfied:

1. Informed consent obtained before any "trial-related activities" (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
2. Diagnosis of plaque psoriasis for at least 6 months with at least one psoriatic plaque measuring between 2 cm and 5 cm at the time of screening
3. If female, subject is either not of childbearing potential (postmenopausal for at least 1 year or surgically sterile) or is of childbearing potential and is using approved method of birth control throughout study and for 1 month after last dose of study drug. Approved methods of birth control include the following:

   1. Condoms, sponge, foams, jellies, diaphragm, or intrauterine device (IUD)
   2. Hormonal contraceptives for 90 days prior to study drug administration
   3. A vasectomized partner
4. Subject must be able and willing to provide written informed consent and comply with requirements of this study protocol

   Following Eligibility & Consent:
5. Subject must be able to donate 130 ml to 490 ml of blood for NKMax America to obtain an adequate number of autologous NK cells necessary to establish the final investigational product
6. Successful establishment of the final NK product, or "study therapy", established by NKMax America

Exclusion Criteria:

Subjects who fulfill any of the following criteria will not be recruited into the study:

1. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
2. Subject has Netherton's syndrome or other genodermatoses that results in a defective epidermal barrier
3. Subjects who have applied topical medication (prescription or over-the-counter) for the treatment of psoriasis to their body within 7 days of the baseline visit
4. Subjects who have taken cyclosporine, methotrexate, immuran, oral retinoids, chemotherapeutic agents, anti-inflammatory biologics (e.g., alefacept, etanercept, etc.), or oral calcineurin inhibitors within 28 days of the whole blood donation visit for the establishment of the investigational product
5. Subjects who are unable to hold their current psoriasis medications for the period of time indicated (at least 7 days for topical medications, at least 28 days for oral or injectable medications) without significant worsening of their psoriasis
6. Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome) or subjects with a history of malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history
7. Subjects receiving phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA]) within 28 days of the baseline visit.
8. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
9. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
10. Subjects with an active bacterial, viral or fungal skin infection (excluding nail fungus)
11. Ongoing participation in an investigational drug trial
12. Presence of psoriasis with exfoliative erythroderma or presence of guttate psoriasis, primary palmoplantar psoriasis, or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for safety is the dose-limiting toxicity (DLT) | From enrollment to end of treatment at 8 Weeks
  DLT is a TEAE of grade ≥3 considered related to SNK01

SECONDARY OUTCOMES:
Preliminary Efficacy by Physician Global Assessment (PGA) | From enrollment to end of treatment at 8 Weeks
  The Physician Global Assessment (PGA) is a 6-point scoring system used to assess disease severity at a given time point. The PGA is a six-point score that summarizes the overall quality (erythema, scaling and thickness) and extent of Psoriasis plaques where (0) is clear, (1) minimal, (2) mild, (3) moderate, (4) severe, and (5) being very severe psoriasis. Change in score from baseline through Week 8 will be assessed.
Preliminary Efficacy by Psoriasis Area and Severity Index (PASI) | From enrollment to end of treatment at 8 Weeks
  Psoriasis Area and Severity Index (PASI) is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). Change in score from baseline through Week 8 will be assessed.
Secondary Safety Measures: Other Non-DLT Adverse Events | From enrollment to end of treatment at 8 Weeks
  Frequency and type of Non-DLT adverse events (graded according to National Cancer Institute's Common Toxicity Criteria for Adverse Events [NCI-CTCAE v 5.0]),

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gutiérrez, MD, Principal Investigator — Hospital Angeles Tijuana
Locations (1):
- Hospital Angeles, Tijuana, Estado de Baja California, Mexico